CLINICAL TRIAL: NCT06585527
Title: A Clinical Study of the Safety and Efficacy of Third-generation Oncolytic TS-2021 in the Treatment of Recurrent Malignant Gliomas
Brief Title: Clinical Study on the Safety and Efficacy of TS-2021 in the Treatment of Recurrent Malignant Glioma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing Neurosurgical Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-1-1071
Record Dates: First submitted 2024-09-03; First posted 2024-09-05 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-07

CONDITIONS: Glioblastoma Multiforme; Glioma, Malignant
Keywords: Oncolytic Virus; Adenovirus; Glioblastoma Multiforme; Glioma, Malignant; Ki-67; TGF-β2; IL-15
MeSH Terms: conditions — Glioblastoma; Glioma; Adenoviridae Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- TS-2021 (Experimental): 30 eligible participants with recurrent malignant glioma will be intratumoral injected the TS-2021 oncolytic virus to study its safety and efficacy.
  Interventions: Biological: TS-2021

INTERVENTIONS:
Biological: TS-2021 — The participants meeting the criteria will undergo TS-2021 oncolytic virus (5×1011PFU/ml) intratumoral injection using stereotactic technique under MR Localization.

SUMMARY:
The goal of this clinical trial is to evaluate the safety and efficacy of oncolytic virus TS-2021 in the treatment of recurrent malignant glioma.About 30 eligible participants with recurrent malignant glioma will :

* Be intratumoral injected the TS-2021 oncolytic virus to study its safety and efficacy.
* Be followed for 1 year after the injection to complete imaging studies, neurological function tests, and report adverse events.

Using the data obtained during the follow-up period, researchers will conduct statistical analyses and evaluate the safety and efficacy of oncolytic virus TS-2021.

ELIGIBILITY:
Inclusion Criteria:

* The patient signed the informed consent voluntarily.
* Age ≥18 years and ≤65 years, male or female.
* After the initial surgery, the imaging showed that the tumor was completely removed, followed by conventional radiotherapy or (and) chemotherapy, and no recurrence was observed within two months after the end of radiotherapy. The patient had a recurrence of supratentorial high-grade glioma. The pathological diagnosis was glioblastoma, anaplastic astrocytoma, anaplastic oligodendroglioma, anaplastic oligodendro-astrocytoma, or subtentorial astrocytoma recurrence.
* After conventional surgery, radiotherapy (or) chemotherapy was performed, and there was no recurrence at the primary site of the tumor, but there was tumor recurrence at the distant site.
* With PET/MRS, tumor recurrence was considered, and the enhanced lesion diameter was greater than 1cm, but less than 3cm.
* KPS score ≥70 before treatment.
* Normal bone marrow reserve function and normal liver and kidney function: Neutrophil absolute value ≥ 1,500/mm3, hemoglobin ≥10 g/dL, platelet count ≥100,000/mm3, total bilirubin level ≤1.5×ULN, glutamic pyruvic transaminase/glutamic oxalacetic transaminase ≤ 2.5× ULN, serum creatinine ≤1.5×ULN, The heart function was normal and the follow-up compliance was good.
* Women of childbearing age (15 to 49 years) must undergo a pregnancy test within 7 days before starting treatment and the result is negative; Fertile men and women must consent to the use of effective contraception to ensure that they do not become pregnant during the study period and for 3 months after stopping treatment.

Exclusion Criteria:

* Pregnant or lactating patients.
* Patients with encephalitis disease, multiple sclerosis, or other CNS (Central Nervous System) infection.
* Patients with a history of organ transplantation or waiting for organ transplantation.
* Patients with uncontrolled infectious diseases or other serious diseases, such as HIV positive.
* Patients with any unstable systemic illness (including active infection, uncontrolled hypertension, unstable angina pectoris, angina pectoris beginning within the last 3 months, congestive heart failure, myocardial infarction occurring within 12 months before enrollment, severe arrhythmia requiring medical treatment, liver or kidney failure, etc.)
* Patients with systemic autoimmune diseases or immunodeficiency diseases.
* Patients with severe allergic constitution.
* Patients with chronic diseases requiring long-term treatment with immune agents or glucocorticoids.
* Patients with mental disorders.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-08-29 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events. | Up to 8 weeks
  All events with a Grade 3 or above toxicity (defined by the CTCAE v4.0) will be tabulated by event and by relationship to TS-2021.
Overall survival | Up to 12 months
  The overall survival for each patient receiving TS-2021 will be calculated.

SECONDARY OUTCOMES:
Objective response rate (ORR) determined by MRI scan review. | Up to 12 months
  Interval tumor size change will be measured.
Progression Free Survival. | Up to 12 months
  Time after TS-2021 administration to clinical and radiographic disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Fusheng Liu, MD,PhD, Study Director — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No